CLINICAL TRIAL: NCT00854451
Title: Relation of Metabolic Rate of Omeprazole and Eradication of Helicobacter Pylori Infection - A Combination of Clinical and Pharmacogenetic Study
Brief Title: Relation of Metabolic Rate of Omeprazole and Eradication of Helicobacter Pylori Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSC86-2314-B002-169
Record Dates: First submitted 2009-02-06; First posted 2009-03-03 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 1996-07

CONDITIONS: Duodenal Ulcer; Helicobacter Pylori Infection
Keywords: Helicobacter pylori; CYP2C19 genotype; intragastric pH; dual therapy; antibiotic resistance
MeSH Terms: conditions — Duodenal Ulcer | interventions — Omeprazole; Amoxicillin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 omeprazole plus amoxicillin (Active Comparator): omeprazole 20mg bid 2wk + amoxicillin 500mg qid 2wk
  Interventions: Drug: omeprazole plus amoxicillin
- 2 omeprazole plus amoxicillin (Active Comparator): omeprazole 20mg bid 2wk + amoxicillin 250mg qid 2wk
  Interventions: Drug: omeprazole plus amoxicillin
- 3 omeprazole plus amoxicillin (Active Comparator): omeprazole 20mg qd 2wk + amoxicillin 500mg qid 2wk
  Interventions: Drug: omeprazole plus amoxicillin
- 4 omeprazole plus amoxicillin (Active Comparator): omeprazole 20mg qd 2wk + amoxicillin 250mg qid 2wk
  Interventions: Drug: omeprazole plus amoxicillin

INTERVENTIONS:
Drug: omeprazole plus amoxicillin
  Arms: 1 omeprazole plus amoxicillin
Drug: omeprazole plus amoxicillin
  Arms: 2 omeprazole plus amoxicillin
Drug: omeprazole plus amoxicillin
  Arms: 3 omeprazole plus amoxicillin
Drug: omeprazole plus amoxicillin
  Arms: 4 omeprazole plus amoxicillin

SUMMARY:
The aims of this study are (1) to evaluate the prevalence rate of PM of CYP2C19 in our country; (2) to evaluate the efficacy of dual therapy with different dose of omeprazole and amoxicillin; (3) to judge the relationship of genotype of CYP2C19 and the eradication rate of dual therapy in the peptic ulcer patients; (4) to try to find out a predictor of success of dual therapy and an optimal dose of dual therapy as first-line and rescue anti-Helicobacter pylori regimen.

DETAILED DESCRIPTION:
Anti-H. pylori therapy is now recommended in patients with peptic ulcer disease associated with bacterial infection. Dual therapy containing one PPI and amoxicillin has been suggested to be a better treatment than classical triple therapy containing bismuth, metronidazole, and tetracycline for H. pylori eradication due to its better compliance and fewer side effects. However, the variation in the eradication rate among different studies has limited its clinical application. Nonetheless, the amoxicillin-based dual therapy, with very rare prevalence of primary and secondary antibiotic resistance, has the potential to be an optimal first-line and rescue anti-Helicobacter pylori regimen if the confounding factors that cause the labile treatment outcome can be clarified. Cytochrome P450 2C19(CYP2C19), the enzyme that metabolizes omeprazole, was found to have genetic polymorphism in its enzyme activity. The percentage of poor metabolizer(PM) of CYP2C19 was much higher in Oriental(18~23%) comparing to Caucasian(3~5%).

The aims of this study is to try to find out a predictor of success of dual therapy and an optimal dose of dual therapy as first-line and rescue anti-Helicobacter pylori regimen. About 130 patients with Hp positive duodenal ulcer will be enrolled and allocated randomly into one of four treatment groups:Group A：omeprazole 20mg bid 2wk + amoxicillin 500mg qid 2wk; Group B：omeprazole 20mg bid 2wk + amoxicillin 250mg qid 2wk; Group C：omeprazole 20mg qd 2wk + amoxicillin 500mg qid 2wk; Group D：omeprazole 20mg qd 2wk + amoxicillin 250mg qid 2wk. All patients will receive endoscopic exam with biopsy again within 1~2 months after the end of treatment. The status of H. pylori infection was examined by endoscopy or the 13C-urea breath test (if the patients refused the second endoscopy). Biopsy from the antrum and body will be taken for the culture, histology and CLO test. Twenty-four hours intragastric pH measurements will be performed on 6 randomly selective patients of each group when these patients complete the first week course of treatment. PCR-RFLP method will be used to detect genotype of CYP2C19 polymorphism using the genomic DNA extracted from the whole blood in all 130 treated patients. The genotyping results will be correlated with the H. pylori eradication rate and intragastric pH value.

The equivalence of demographic information among various treatment groups or genotypes will be revealed by chi-square independence test, t-test, one-way ANOVA, or Kruskal-Wallis test. The above statistical methods as well as Mann-Whitney test will be also used to analyze clinical outcome. Confidence intervals for eradication rates will be computed by plus-four method. Multiple logistic regression will be used to explore the predictor of the eradication outcome. Multiple regression will be used to explore the predictor of the intragastric acidity. A p-value less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Male and female dyspeptic patients with H. pylori-positive duodenal ulcer.

Exclusion Criteria:

* Pregnant or nursing woman
* Serious concomitant illness
* Malignant tumor of any kind
* Serious bleeding during the course of this ulcer
* Previous gastric surgery
* Taking bismuth compounds, proton pump inhibitors, antibiotic or non-steroid anti-inflammatory drugs for at least one month prior to pretreatment endoscopy.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 1996-08; Primary Completion 1997-12 (Actual); Study Completion 1998-02 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate and intragastric pH value

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Chin Yang, M.D., Principal Investigator — Department of Internal Medicine, National Taiwan University Hospital
Locations (1):
- Department of Internal Medicine, National Taiwan University Hospital, Taipei, Taiwan